CLINICAL TRIAL: NCT04976881
Title: Promoting Preconception Care and Diabetes Self-Management Among Reproductive-Aged Women With Diabetes: The PREPARED Trial
Brief Title: Promoting Preconception Care and Diabetes Self-Management Among Reproductive-Aged Women With Diabetes
Acronym: PREPARED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other); AllianceChicago (Other)
Responsible Party: Principal Investigator, Stacy C Bailey, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: STU00214604
Record Dates: First submitted 2021-07-15; First posted 2021-07-26 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Diabetes Mellitus, Type 2; Electronic Health Record; Primary Health Care; Reproductive Behavior
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Reproductive Behavior | interventions — Medication Reconciliation; Equipment and Supplies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Care (No Intervention): Usual care includes: 1) no specific materials to promote medication reconciliation, reproductive planning, or patient education on diabetes self-management within the context of preconception care, 2) variable physician preconception counseling without any EHR notifications or counseling support; and 3) no specific patient support or prompts to promote healthy behaviors post-visits.
- PREPARED Strategy (Active Comparator): Our PREPARED strategy will utilize health information and consumer technologies to 'hardwire' preconception care and promote diabetes self-management among reproductive-aged, adult women with T2DM in primary care. PREPARED will leverage electronic health record technology at clinic visits to: [1] promote medication reconciliation and safety, [2] prompt provider preconception counseling, and [3] deliver low literacy print tools to reinforce counseling and promote diabetes self-care. Post-visit, text messaging will be used to: [4] encourage healthy lifestyle behaviors.
  Interventions: Behavioral: Medication Reconciliation (MedRec) Tool; Behavioral: Provider Alert and Decision Support; Behavioral: PREPSheet; Behavioral: Text Messaging

INTERVENTIONS:
Behavioral: Medication Reconciliation (MedRec) Tool — Patients will receive a print MedRec tool, generated via the EHR, which includes a list of medications prescribed according to the patient record. Patients are asked to review this list, to add/remove drugs to reflect actual use, to note how they are taking each medication, and to describe any concerns.
  Arms: PREPARED Strategy
Behavioral: Provider Alert and Decision Support — During the clinic visit, an automated, EHR alert will notify the provider that the patient is a woman of reproductive age with T2DM and should receive counseling on the importance of glycemic control, the use of contraception until glycemic control is achieved, and the benefits of folic acid.
  Arms: PREPARED Strategy
Behavioral: PREPSheet — When patients leave an encounter, they will receive a patient-friendly educational material (a.k.a. the PREPSheet) that reviews potential risks of pregnancy in the context of T2DM and highlights the importance of: 1) achieving glycemic control through diabetes self-care, 2) using effective contraception until glycemic control is achieved and pregnancy is desired, 3) discussing medication use with a provider if planning or becoming pregnant, and 4) taking folic acid daily to reduce increased risk of neural tube defects.
  Arms: PREPARED Strategy
Behavioral: Text Messaging — Within ~5 days of their index clinic visit, intervention patients will begin to receive daily, unidirectional text messages to reinforce diabetes self-care behaviors.
  Arms: PREPARED Strategy

SUMMARY:
This study is being done to investigate strategies that may improve patient's knowledge of type 2 diabetes during reproductive age and improve knowledge and engagement in self-care activities.

DETAILED DESCRIPTION:
Our Promoting REproductive Planning, And REadiness in Diabetes (PREPARED) strategy will utilize health information and consumer technologies to 'hardwire' preconception care and promote diabetes self-management among reproductive-aged, adult women with T2DM in primary care. Specifically, PREPARED will leverage electronic health record (EHR) technology at clinic visits to: [1] promote medication reconciliation and safety, [2] prompt patient-provider preconception counseling and reproductive planning, and [3] deliver low literacy print tools to reinforce counseling and promote goal-setting for diabetes self-care activities. Post-visit, a widely-available text messaging platforms will be used to: [4] encourage healthy lifestyle behaviors through goal-setting and daily reminders. Our randomized trial will assess the effectiveness and fidelity of a technology-based strategy to promote preconception care and diabetes self-management among women with type 2 diabetes in primary care.

Aim 1: Test the effectiveness of PREPARED, compared to usual care, to improve patient: a) knowledge of reproductive risks associated with T2DM and recommended self-care activities b) engagement in self-care behaviors, including: i) diet, ii) physical activity, iii) adherence to diabetes medications; and use of iv) folic acid, and v) most or moderately effective contraception, when indicated; and c) clinical measures, including hemoglobin A1c, blood pressure, and LDL cholesterol.

Aim 2: Assess whether PREPARED reduces disparities in the above outcomes versus usual care.

Aim 3: Evaluate the fidelity of PREPARED to prompt medication reconciliation and preconception counseling, and to deliver patient education and post-visit support of diabetes self-care behaviors.

ELIGIBILITY:
Inclusion Criteria:

* female
* age 18-44
* English or Spanish-speaking
* have a chart diagnosis of type 2 diabetes
* not currently pregnant
* not infecund, sterilized, or in a monogamous relationship with a sterilized partner
* have a private cell phone with text messaging capability.

Exclusion Criteria:

* severe, uncorrectable vision, hearing, or cognitive impairments that would preclude study consent or participation

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 840 (Estimated)
Dates: Start 2022-05-06 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Average difference in HbA1c values between Intervention and Control Patients | 6 months
  We will abstract HbA1c values from performance sites EHRs to investigate effects of PREPARED.
Knowledge of reproductive risks | 1 month
  We will use a questionnaire, developed by our team and the scientific literature, to evaluate patient knowledge of reproductive risks and recommended health behaviors for women with type 2 diabetes. It includes items assessing knowledge of pregnancy planning, reproductive risks, and desired diabetes self-care behaviors. Correctly answered questions will be summed and a total knowledge score will be generated. Higher scores indicate greater knowledge.

SECONDARY OUTCOMES:
Average difference in blood pressure values between Intervention and Control Patients | 6 months
  We will abstract blood pressure values (systolic and diastolic) from performance sites EHRs to investigate effects of PREPARED.
Average difference in cholesterol values between Intervention and Control Patients | 6 months
  We will abstract cholesterol values from performance sites EHRs to investigate effects of PREPARED.
Engagement in diabetes self-care activities | at 1 month and 3 months
  We will use the validated Summary of Diabetes Self Care Activities (SDSCA) measure. Scores range from 0 to 7 for each domain, with higher scores reflect greater engagement.
Contraceptive use | at 1 month and 3 months
  we will use validated items to assess patient contraceptive use, which is categorized into use of a 'most or moderately effective' form of contraception or 'less effective/no contraception'
Folic acid use | at 1 month and 3 months
  Patients are asked if they have taken folic acid supplements or a vitamin containing folic acid over the past month (yes/no).

CONTACTS AND LOCATIONS:
Overall Officials: Stacy Bailey, PhD MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon reasonable request to the study principal investigator.
Supporting Information: Study Protocol, ICF
Time Frame: Data and other documents will be made available upon reasonable request to the PI 24 months after study termination

REFERENCES:
- [Derived] Bailey SC, Pack AP, Wismer G, Calderon N, Velazquez E, Batio S, Ekong A, Eggleston A, Wallia A, Wolf MS, Schauer JM, Tenfelde S, Liebovitz DM, Grobman WA. Promoting REproductive Planning And REadiness in Diabetes (PREPARED) Study protocol: a clinic-randomised controlled trial testing a technology-based strategy to promote preconception care for women with type 2 diabetes. BMJ Open. 2023 Nov 8;13(11):e078282. doi: 10.1136/bmjopen-2023-078282. PMID 37940161

DOCUMENTS (1):
  • Informed Consent Form (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/81/NCT04976881/ICF_000.pdf